CLINICAL TRIAL: NCT01807130
Title: Automated MEdical Record Driven Implantable CArdioverter-defibrillator Heart Failure Trial (AMERICA-HF)
Acronym: AMERICA-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We observed a very high referral rate for patients with HF in the Duke Health System, eliminating the need for an automated referral process.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00042120
Record Dates: First submitted 2013-03-05; First posted 2013-03-08 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-08

CONDITIONS: Heart Failure
Keywords: Heart Failure; Medical Therapy; ICD; CRT
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Registry (Placebo Comparator): Patients randomized to the registry arm will be followed per usual standard of care by their primary providers. Those providers may refer to subspecialty HF or electrophysiology care as they see fit.
  Interventions: Other: Placebo (Registry Arm)
- Intervention (Experimental): Patients in the intervention arm without compelling contraindications to HF therapies will be referred automatically to specialists in HF or electrophysiology with recommendations to consider those therapies that are not in compliance with guidelines.
  Interventions: Other: Automated HF/EP Referral

INTERVENTIONS:
Other: Automated HF/EP Referral — Patients in the intervention arm without compelling contraindications to HF therapies will be referred automatically to specialists in HF or electrophysiology (EP) with recommendations to consider those therapies that are not in compliance with guidelines.
  Arms: Intervention
Other: Placebo (Registry Arm) — Patients assigned to the registry will receive referral to specialists in HF or EP as deemed necessary by the patients physicians.
  Arms: Registry

SUMMARY:
Purpose and Objective: Heart failure therapies including beta-blockers, ACE-inhibitors, aldosterone antagonists, implantable cardioverter-defibrillator (ICD) and cardiac resynchronization therapy (CRT) devices have proven beneficial but are underused in eligible patients. The investigators seek to determine if automating referral to cardiologists and electrophysiologists through an intelligent electronic medical record system can improve adherence to American College of Cardiology (ACC)/ American Heart Association (AHA) heart failure guideline recommended therapies.

Study activities and population group: The AMERICA-HF trial will be a randomized, single-center, single blinded study comparing standard-practice provider initiated cardiovascular specialty referral to experimental automated medical record driven cardiovascular specialty referral. An investigational program will automatically screen all finalized electronic reports from clinically indicated transthoracic echocardiogram studies performed in the Duke University Echo Lab system and create an automated query to obtain HF ICD-9 codes. Eligible patients will be randomly assigned to participate in a registry (n=125) or automated electronic medical record (EMR) based subspecialty care intervention arm (n=125).

Data analysis: The primary endpoint is rate of adherence (%) to ACC/AHA HF guideline recommended therapies at 3, 6, and 12 month follow-up among patients randomized to the registry compared to the intervention. Differences in characteristics (including use of guideline recommended therapies) will be tested using Pearson Chi-square tests for categorical variables and Wilcoxon two-sample tests for continuous variables. Time to event analysis will be performed for the secondary endpoints of hospitalization or death.

ELIGIBILITY:
Inclusion Criteria:

* Left Ventricular Ejection Fraction ≤ 35% on transthoracic echocardiogram
* One of the following ICD-9 HF diagnostic codes 398.91, 428.0, 428.1, 428.2x, 428.3x, 428.4x, 428.9

Exclusion Criteria:

* Pregnancy
* Inability to speak English
* Inability to provide verbal consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Rate of adherence (%) to ACC/AHA HF guideline recommended HF therapies among patients randomized to the registry compared to the intervention | 12 month follow-up

SECONDARY OUTCOMES:
Adherence to ACC/AHA guideline recommended therapies by sex and race compared to standard referral processes among patients with ejection fraction (EF) ≤ 35% and symptomatic HF. | 12 months
Repeated Measures Analysis of Adherence to ACC/AHA HF Guidelines | 3, 6, 12 months
  To determine the time-frame over which the intervention has a treatment effect, repeated measures analysis will be performed at 3 months, 6 months, and 12 months after the intervention is made. The goal of this analysis to to determine how quickly adherence is achieved with the intervention and whether adherence is maintained long-term.

CONTACTS AND LOCATIONS:
Overall Officials: Brett D Atwater, MD, Principal Investigator — Duke University; Jason I Koontz, MD/PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States